CLINICAL TRIAL: NCT01073605
Title: A Two Years Multicentre Study of Genotropin Treatment of Short Prepubertal Children With Intra-Uterine Growth Retardation
Brief Title: Genotropin Treatment in Short Prepubertal Children With Intra-Uterine Growth Retardation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 93-8122-001; A6281186, CTN 93-8122-001
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Results first posted 2010-08-31 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-02

CONDITIONS: Growth Disorders; Intrauterine Growth Retardation
Keywords: Short height; intra-uterine growth retardation; Genotonorm; continuous treatment; intermittent treatment
MeSH Terms: conditions — Growth Disorders; Fetal Growth Retardation | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Genotonorm A (Active Comparator): Continuous 0.7 IU/kg/week or 0.03 mg/kg/day
  Interventions: Drug: Genotonorm
- Genotonorm B (Active Comparator): Continuous, 1.4 IU/kg/week or 0.06 mg/kg/day
  Interventions: Drug: Genotonorm
- Genotonorm C (Active Comparator): Intermittent, 1.4 IU/kg/week or 0.06 mg/kg/day
  Interventions: Drug: Genotonorm

INTERVENTIONS:
Drug: Genotonorm — 0.7 IU/kg/week or 0.03 mg/kg/day, daily subcutaneous injection
  Arms: Genotonorm A
Drug: Genotonorm — 1.4 IU/kg/week or 0.06 mg/kg/day, daily subcutaneous injection
  Arms: Genotonorm B
Drug: Genotonorm — 1.4 IU/kg/week or 0.06 mg/kg/day, daily subcutaneous injection Intermittent treatment (6 months with treatment and 6 months without)
  Arms: Genotonorm C

SUMMARY:
To evaluate the effect of continuous and intermittent administration of Genotonorm on stature in short prepubertal children with intra-uterine growth retardation

ELIGIBILITY:
Inclusion Criteria:

* Chronological age (CA) between 3 and 10 for girls
* Chronological age between 3 and 12 for boys
* Height for CA below - 2 SD
* Birth length for CA below -2SD

Exclusion Criteria:

* Endocrine disease except well-substituted hypothyroidism
* Sever chronic disease
* Skeletal dysplasia
* Known chromosomal aberration
* Ongoing treatment with steroids
* Known intrauterine infection

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 1993-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- France (28):
  - Pfizer Investigational Site, Angers, France
  - Pfizer Investigational Site, Grenoble, France
  - Pfizer Investigational Site, Paris, France
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Boulogne
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Bron
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Hyères
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Reims
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Saint-Priest-en-Jarez
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Tarbes
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Tours
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=93-8122-001&StudyName=Genotropin%20Treatment%20in%20Short%20Prepubertal%20Children%20with%20Intra-Uterine%20Growth%20Retardation

RESULTS

PARTICIPANT FLOW:
Groups:
- Genotonorm 0.7 (Continuous Treatment): Subjects received 0.7 international unit (IU)/kilogram (kg)/week (0.03 milligram [mg]/kg/day) of Genotonorm growth hormone (GH) as a continuous treatment. Treatment was allowed to be taken until final height of the subject had been reached.
- Genotonorm 1.4 (Continuous Treatment): Subjects received 1.4 IU/kg/week (0.06 mg/kg/day) of the growth hormone Genotonorm as a continuous treatment. Treatment was allowed to be taken until final height of the subject had been reached.
- Genotonorm 1.4 (Intermittent Treatment): Subjects received 1.4 IU/kg/week (0.06 mg/kg/day) of the growth hormone Genotonorm as an intermittent treatment. Treatment was allowed to be taken until final height of the subject had been reached.
Period: Overall Study
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Started | 68 | 71 | 69
Received Treatment | 68 | 70 | 68
Completed | 6 (Corresponds to follow-up until final height) | 4 (Corresponds to follow-up until final height) | 8 (Corresponds to follow-up until final height)
Not Completed | 62 | 67 | 61
Not completed — Ongoing at Cutoff Date | 1 | 1 | 0
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Lost to Follow-up | 3 | 4 | 9
Not completed — Other | 25 | 21 | 29
Not completed — Withdrawal by Subject | 31 | 39 | 22
Not completed — Randomized But Not Treated | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Genotonorm 0.7 (Continuous Treatment): Subjects received 0.7 IU/kg/week (0.03 mg/kg/day) of the growth hormone Genotonorm as a continuous treatment. Treatment was allowed to be taken until final height of the subject had been reached.
- Total: Total of all reporting groups
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment) | Total
Number analyzed (Participants) | 68 | 70 | 68 | 206
Age, Customized [Number; unit: Participants]
  < 4 years | 15 | 8 | 6 | 29
  4 - 8 years | 29 | 32 | 29 | 90
  8 - 12 years | 23 | 30 | 33 | 86
  >= 12 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 31 | 39 | 95
  Male | 43 | 39 | 29 | 111

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Annual Growth Rate Measured at 2 Years Following Treatment With Genotonorm
Description: Annual growth rate was expressed as height velocity (centimeter [cm]/year). This was derived by substracting annual growth rate at Baseline from 2-year value. (Annual growth rate was calculated each year and rescaled to 1 year if the interval between x and x-1 was not 365 days, as long as a subject remains in the study): ANGRYx = (Height Yx - Height Y{x-1}) / {(Date of Yx - Date of Y{x-1}) /365.25}
Time Frame: Baseline, 2 years
Population: All subjects who received at least 1 study dose of Genotonorm were included in the Full Analysis Set (FAS). Number of Participants Analyzed = number of subjects with change in annual growth rate at 2 years.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 47 | 37 | 40
cm/year | 3.07 (2.21) | 3.97 (1.72) | 2.84 (1.71)
Statistical Analysis 1: Comparison: Genotonorm 0.7 (Continuous Treatment) vs Genotonorm 1.4 (Continuous Treatment); Test type: Superiority or Other; p = 0.02922, Wilcoxon (Mann-Whitney) — P-values for the 3 treatment comparisons should be interpreted in line with the Bonferroni stepwise (Holm) testing procedure, to maintain the Type 1 error at p=0.05
Statistical Analysis 2: Comparison: Genotonorm 0.7 (Continuous Treatment) vs Genotonorm 1.4 (Intermittent Treatment); Test type: Superiority or Other; p = 0.74299, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Genotonorm 1.4 (Continuous Treatment) vs Genotonorm 1.4 (Intermittent Treatment); Test type: Superiority or Other; p = 0.00467, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Annual Growth Rate Standard Deviation Score (SDS)
Description: Calculated using Sempe reference means and standard deviations for growth rate according to age and sex. Standardization was performed for chronological age.
Time Frame: Baseline, 1 to 6 years
Population: FAS. Number of Participants Analyzed = number of subjects with evaluable data at Baseline. n = number of subjects with evaluable data at each time point. Data beyond 6 years are not reported due to the low proportion of subjects followed up beyond 6 years.
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 50 | 42 | 43
SDS
  Baseline (n=50, 42, 43) | -2.72 (1.83) | -2.58 (1.39) | -2.75 (1.73)
  1 year (n=57, 55, 59) | 2.14 (1.52) | 3.97 (2.26) | 1.71 (1.51)
  2 years (n=53, 49, 56) | 0.77 (1.57) | 2.00 (1.73) | 0.67 (1.22)
  3 years (n=39, 34, 41) | 0.36 (1.14) | 1.35 (1.78) | 0.31 (1.12)
  4 years (n=21, 18, 27) | 0.13 (1.55) | 0.61 (1.20) | 0.34 (1.20)
  5 years (n=12, 10, 20) | 0.18 (1.24) | 0.09 (0.88) | -0.02 (1.46)
  6 years (n=11, 7, 19) | 0.90 (1.92) | 0.59 (1.61) | 0.05 (1.20)

3. Secondary Outcome: Change From Baseline in Annual Growth Rate SDS
Description: Calculated corresponding to the gender and chronological age by substracting annual growth rate SDS at Baseline from annual growth rate SDS at each year.
Time Frame: Baseline, 1 to 3 years
Population: FAS. Number of Participants Analyzed = number of subjects with evaluable data at 1 year. n = number of subjects with evaluable data at each time point.
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 49 | 42 | 42
SDS
  1 year (n=49, 42, 42) | 4.81 (2.27) | 6.56 (2.55) | 4.37 (2.16)
  2 years (n=47, 37, 40) | 3.51 (2.50) | 4.53 (1.89) | 3.37 (2.33)
  3 years (n=34, 25, 32) | 3.31 (2.06) | 3.80 (2.20) | 3.17 (1.86)
Statistical Analysis 1: Comparison: Genotonorm 0.7 (Continuous Treatment) vs Genotonorm 1.4 (Continuous Treatment); 1 year; Test type: Superiority or Other; p = 0.00125, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Genotonorm 0.7 (Continuous Treatment) vs Genotonorm 1.4 (Intermittent Treatment); 1 year; Test type: Superiority or Other; p = 0.25995, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Genotonorm 1.4 (Continuous Treatment) vs Genotonorm 1.4 (Intermittent Treatment); 1 year; Test type: Superiority or Other; p = 0.00008, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Genotonorm 0.7 (Continuous Treatment) vs Genotonorm 1.4 (Continuous Treatment); 2 years; Test type: Superiority or Other; p = 0.03273, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Genotonorm 0.7 (Continuous Treatment) vs Genotonorm 1.4 (Intermittent Treatment); 2 years; Test type: Superiority or Other; p = 0.68581, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Genotonorm 1.4 (Continuous Treatment) vs Genotonorm 1.4 (Intermittent Treatment); 2 years; Test type: Superiority or Other; p = 0.00530, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Genotonorm 0.7 (Continuous Treatment) vs Genotonorm 1.4 (Continuous Treatment); 3 years; Test type: Superiority or Other; p = 0.57556, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Genotonorm 0.7 (Continuous Treatment) vs Genotonorm 1.4 (Intermittent Treatment); 3 years; Test type: Superiority or Other; p = 0.63956, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Genotonorm 1.4 (Continuous Treatment) vs Genotonorm 1.4 (Intermittent Treatment); 3 years; Test type: Superiority or Other; p = 0.16421, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Height (cm)
Description: Performed by use of a wallmounted device (eg, Harpenden Stadiometer). Each subject was measured 3 times and the mean of these measurements was recorded as the present height. Final Height: Children are defined as reaching their final height when annual Growth Rate is less than 2 cm in the previous year and bone age is equal to or greater than 17 years in boys and equal to or greater than 15 years in girls.
Time Frame: Baseline, 1 to 6 years, final height
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 58 | 56 | 60
cm
  Baseline (n=58, 56, 60) | 105.22 (15.04) | 107.06 (12.29) | 106.44 (12.04)
  1 year (n=57, 55, 59) | 113.38 (15.09) | 116.31 (12.24) | 113.71 (12.01)
  2 years (n=53, 49, 56) | 119.67 (15.18) | 124.11 (13.02) | 120.64 (12.34)
  3 years (n=39, 34, 41) | 123.92 (15.08) | 131.75 (13.76) | 125.39 (12.52)
  4 years (n=21, 18, 27) | 124.67 (13.14) | 132.30 (13.23) | 127.59 (11.51)
  5 years (n=12, 10, 21) | 126.73 (10.01) | 131.01 (9.26) | 129.98 (9.93)
  6 years (n=11, 7, 20) | 133.29 (10.46) | 138.84 (8.69) | 135.45 (10.10)
  Final height (n=17, 12, 22) | 146.86 (11.26) | 151.98 (6.52) | 149.13 (9.07)

5. Secondary Outcome: Change From Baseline in Height (cm)
Description: Calculated by substracting height at Baseline from height at each year. Final Height: Children are defined as reaching their final height when annual Growth Rate is less than 2 cm in the previous year and bone age is equal to or greater than 17 years in boys and equal to or greater than 15 years in girls.
Time Frame: Baseline, 1 to 6 years, final height
Population: FAS. Number of Participants Analyzed = number of subjects with evaluable data at Baseline. n = number of subjects with evaluable data at Baseline and each time point. Data beyond 6 years are not reported due to the low proportion of subjects followed up beyond 6 years.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 58 | 56 | 60
cm
  1 year (n=57, 55, 59) | 8.21 (1.38) | 9.21 (1.45) | 7.33 (1.32)
  2 years (n=53, 49, 56) | 14.77 (2.45) | 17.01 (2.21) | 13.92 (2.03)
  3 years (n=39, 34, 41) | 20.62 (3.00) | 24.49 (3.04) | 20.14 (2.78)
  4 years (n=21, 18, 27) | 26.36 (4.37) | 30.77 (3.43) | 25.83 (3.26)
  5 years (n=12, 10, 21) | 32.23 (5.92) | 35.70 (4.27) | 32.16 (3.81)
  6 years (n=11, 7, 20) | 38.20 (6.66) | 44.03 (3.09) | 38.01 (4.82)
  Final height (n=17, 12, 22) | 45.39 (13.08) | 45.30 (13.72) | 40.93 (9.22)

6. Secondary Outcome: Height (SDS)
Description: Calculated using Sempe reference means and standard deviations for height. Final Height: Children are defined as reaching their final height when annual Growth Rate is less than 2 cm in the previous year and bone age is equal to or greater than 17 years in boys and equal to or greater than 15 years in girls.
Time Frame: Baseline, 1 to 6 years, final height
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 58 | 56 | 60
SDS
  Baseline (n=58, 56, 60) | -3.16 (0.52) | -3.07 (0.46) | -3.21 (0.65)
  1 year (n=57, 55, 59) | -2.49 (0.54) | -2.17 (0.50) | -2.68 (0.69)
  2 years (n=53, 49, 56) | -2.21 (0.66) | -1.68 (0.52) | -2.38 (0.75)
  3 years (n=39, 34, 41) | -2.17 (0.70) | -1.38 (0.57) | -2.24 (0.90)
  4 years (n=21, 18, 27) | -2.16 (1.03) | -1.16 (0.73) | -2.09 (0.96)
  5 years (n=12, 10, 21) | -1.95 (1.26) | -1.15 (0.83) | -1.96 (1.10)
  6 years (n=11, 7, 19) | -1.80 (1.28) | -0.67 (0.66) | -1.93 (1.18)
  Final height (n=14, 9, 18) | -2.06 (0.76) | -1.97 (0.95) | -2.29 (1.35)

7. Secondary Outcome: Change From Baseline in Height (SDS)
Description: Calculated by substracting height SDS at Baseline from height SDS at each year. Final Height: Children are defined as reaching their final height when annual Growth Rate is less than 2 cm in the previous year and bone age is equal to or greater than 17 years in boys and equal to or greater than 15 years in girls.
Time Frame: Baseline, 1 to 6 years, final height
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 58 | 56 | 60
SDS
  1 year (n=57, 55, 59) | 0.67 (0.28) | 0.88 (0.30) | 0.53 (0.28)
  2 years (n=53, 49, 56) | 0.94 (0.45) | 1.40 (0.43) | 0.84 (0.37)
  3 years (n=39, 34, 41) | 1.06 (0.54) | 1.70 (0.54) | 0.99 (0.51)
  4 years (n=21, 18, 27) | 1.20 (0.81) | 1.98 (0.69) | 1.21 (0.54)
  5 years (n=12, 10, 21) | 1.37 (1.12) | 2.03 (0.87) | 1.46 (0.69)
  6 years (n=11, 7, 19) | 1.54 (1.12) | 2.60 (0.66) | 1.54 (0.86)
  Final height (n=14, 9, 18) | 1.00 (0.53) | 0.97 (0.95) | 0.86 (1.16)
Statistical Analysis 1: Comparison: Genotonorm 0.7 (Continuous Treatment) vs Genotonorm 1.4 (Continuous Treatment); 3 years; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Genotonorm 0.7 (Continuous Treatment) vs Genotonorm 1.4 (Intermittent Treatment); 3 years; Test type: Superiority or Other; p = 0.58324, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Genotonorm 1.4 (Continuous Treatment) vs Genotonorm 1.4 (Intermittent Treatment); 3 years; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Body Mass Index (BMI)
Description: BMI was calculated by weight divided by height squared.
Time Frame: Baseline, 1 to 6 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 58 | 56 | 60
kg/m^2
  Baseline (n=58, 56, 60) | 14.74 (1.48) | 15.14 (1.76) | 14.59 (1.51)
  1 year (n=56, 55, 59) | 14.82 (1.52) | 15.44 (1.94) | 14.87 (1.76)
  2 years (n=53, 49, 56) | 15.33 (1.78) | 15.92 (2.15) | 15.29 (2.00)
  3 years (n=39, 34, 41) | 15.59 (2.02) | 16.65 (2.92) | 15.58 (2.11)
  4 years (n=21, 18, 27) | 15.32 (1.56) | 17.03 (3.70) | 15.80 (2.37)
  5 years (n=12, 10, 21) | 15.80 (1.57) | 16.25 (1.70) | 16.69 (3.92)
  6 years (n=11, 7, 20) | 16.21 (1.46) | 16.34 (1.80) | 17.28 (4.21)

9. Secondary Outcome: Weight
Time Frame: Baseline, 1 to 6 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 58 | 56 | 60
kg
  Baseline (n=58, 56, 60) | 16.77 (5.43) | 17.70 (5.12) | 16.79 (4.35)
  1 year (n=56, 55, 59) | 19.71 (6.28) | 21.29 (6.04) | 19.56 (5.17)
  2 years (n=53, 49, 56) | 22.66 (7.62) | 25.08 (7.43) | 22.64 (6.05)
  3 years (n=39, 34, 41) | 24.77 (8.80) | 29.61 (9.62) | 24.98 (7.05)
  4 years (n=21, 18, 27) | 24.30 (7.01) | 30.56 (10.42) | 26.28 (7.94)
  5 years (n=12, 10, 21) | 25.74 (6.22) | 28.07 (5.22) | 28.52 (8.96)
  6 years (n=11, 7, 21) | 29.13 (6.42) | 31.94 (7.28) | 32.30 (10.32)

10. Secondary Outcome: Change From Baseline in Bone Age
Description: Bone age was determined by the Greulich-Pyle method. Calculated by substracting bone age at Baseline from bone age at each year
Time Frame: Baseline, 1 to 3 years
Population: Safety population = all subjects who received at least 1 study dose of GH. Number of Participants Analyzed = number of subjects with evaluable data at Baseline. n = number of subjects with evaluable data at Baseline and each time point.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 61 | 62 | 61
Years
  1 year (n=53, 60, 56) | 1.17 (0.51) | 1.27 (0.72) | 1.25 (0.54)
  2 years (n=52, 51, 49) | 2.40 (0.90) | 2.50 (1.08) | 2.58 (0.97)
  3 years (n=41, 39, 35) | 3.53 (1.22) | 4.06 (1.05) | 3.67 (0.97)

11. Secondary Outcome: Change From Baseline in Bone Age/Change From Baseline in Chronological Age Ratio
Description: Bone age was determined by the Greulich-Pyle method. Chronological Age (years) was calculated as: (Date minus Date of Birth) divided by 365.25. Chronological Age used was the age at the date that the corresponding Bone Age X-ray was performed. Ratio was calculated by change from Baseline in bone age divided by change from Baseline in chronological age.
Time Frame: 1 to 3 years
Population: Safety population = all subjects who received at least 1 study dose of GH. Number of Participants Analyzed = number of subjects with evaluable data at 1 year. n = number of subjects with evaluable data at each time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 53 | 60 | 56
ratio
  1 year (n=53, 60, 56) | 0.96 (0.41) | 1.07 (0.62) | 1.06 (0.45)
  2 years (n=51, 51, 49) | 1.06 (0.41) | 1.14 (0.50) | 1.18 (0.44)
  3 years (n=35, 37, 35) | 1.09 (0.39) | 1.26 (0.32) | 1.14 (0.29)

12. Secondary Outcome: Chronological Age at Onset of Puberty
Description: Chronological age (years) at first study visit with onset of puberty = (Date of study visit minus Date of Birth) divided by 365.25.
Time Frame: Onset of puberty
Population: Safety population. Number of participants analyzed = number of subjects who started puberty by the end of the study.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 30 | 35 | 45
Years | 11.88 (2.22) | 11.12 (1.74) | 11.58 (1.42)
Statistical Analysis 1: Comparison: Genotonorm 0.7 (Continuous Treatment) vs Genotonorm 1.4 (Continuous Treatment); Test type: Superiority or Other; p = 0.0681, ANCOVA — There is no adjustment for multiplicity of treatment comparisons; The Analysis of Covariance took into account the patient covariates age and gender; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [-0.05 to 1.39]
Statistical Analysis 2: Comparison: Genotonorm 0.7 (Continuous Treatment) vs Genotonorm 1.4 (Intermittent Treatment); Test type: Superiority or Other; p = 0.8971, ANCOVA — There is no adjustment for multiplicity of treatment comparisons; The Analysis of Covariance took into account the patient covariates age and gender; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.65 to 0.74]
Statistical Analysis 3: Comparison: Genotonorm 1.4 (Continuous Treatment) vs Genotonorm 1.4 (Intermittent Treatment); Test type: Superiority or Other; p = 0.0583, ANCOVA — There is no adjustment for multiplicity of treatment comparisons; The Analysis of Covariance took into account the patient covariates age and gender; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.27 to 0.02]

13. Secondary Outcome: Number of Subjects Reaching Puberty
Description: The defined criteria for reaching puberty were: boy=if right or left testes volume ≥4 ml; girl=if breast development ≥2. Tanner Adolescent Pubertal Staging Questionnaire documents the stage of development of secondary sexual characteristics rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size). Onset of puberty was defined as the visit where the data recorded first met the above criteria for starting puberty.
Time Frame: Baseline, 1 to 6 years
Population: Safety population. Number of Participants Analyzed = number of subjects with evaluable data at Baseline. Data beyond 6 years are not reported due to the low proportion of subjects followed up beyond 6 years. Started = started puberty; Not Started = not started puberty yet as per Tanner scale.
Measure: Number; unit: participants
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Number analyzed (Participants) | 68 | 70 | 68
participants
  Baseline (Female, Not Started) | 25 | 31 | 39
  Baseline (Male, Not Started) | 43 | 39 | 29
  1 year (Female, Not Started) | 24 | 27 | 37
  1 year (Female, Started) | 1 | 3 | 2
  1 year (Male, Not Started) | 36 | 35 | 27
  1 year (Male, Started) | 4 | 3 | 1
  2 years (Female, Not Started) | 20 | 20 | 31
  2 years (Female, Started) | 3 | 7 | 6
  2 years (Male, Not Started) | 31 | 28 | 20
  2 years (Male, Started) | 9 | 7 | 6
  3 years (Female, Not Started) | 16 | 10 | 16
  3 years (Female, Started) | 3 | 9 | 11
  3 years (Male, Not Started) | 19 | 15 | 9
  3 years (Male, Started) | 6 | 7 | 4
  4 years (Female, Not Started) | 10 | 7 | 10
  4 years (Female, Started) | 2 | 5 | 7
  4 years (Male, Not Started) | 10 | 5 | 7
  4 years (Male, Started) | 1 | 2 | 3
  5 years (Female, Not Started) | 5 | 4 | 5
  5 years (Female, Started) | 2 | 3 | 10
  5 years (Male, Not Started) | 6 | 6 | 4
  5 years (Male, Started) | 2 | 1 | 1
  6 years (Female, Not Started) | 3 | 3 | 3
  6 years (Female, Started) | 3 | 2 | 12
  6 years (Male, Not Started) | 5 | 4 | 1
  6 years (Male, Started) | 3 | 1 | 4

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Genotonorm 0.7 (Continuous Treatment) | Genotonorm 1.4 (Continuous Treatment) | Genotonorm 1.4 (Intermittent Treatment)
Serious Adverse Events (participants affected / at risk) | 0/68 | 4/70 | 3/68
Other Adverse Events (participants affected / at risk) | 40/68 | 42/70 | 35/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotonorm 0.7 (Continuous Treatment) (N=68) | Genotonorm 1.4 (Continuous Treatment) (N=70) | Genotonorm 1.4 (Intermittent Treatment) (N=68)
Tonsillectomy (Surgical and medical procedures) | 0 | 4 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Genotonorm 0.7 (Continuous Treatment) (N=68) | Genotonorm 1.4 (Continuous Treatment) (N=70) | Genotonorm 1.4 (Intermittent Treatment) (N=68)
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 4
Pyrexia (General disorders) | 4 | 3 | 3
Bronchitis (Infections and infestations) | 13 | 9 | 17
Ear infection (Infections and infestations) | 15 | 15 | 9
Fungal infection (Infections and infestations) | 4 | 1 | 0
Gastroenteritis (Infections and infestations) | 4 | 8 | 11
Influenza (Infections and infestations) | 6 | 9 | 7
Nasopharyngitis (Infections and infestations) | 16 | 16 | 11
Pharyngitis (Infections and infestations) | 2 | 6 | 7
Rhinitis (Infections and infestations) | 4 | 2 | 6
Tracheitis (Infections and infestations) | 3 | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 19 | 19 | 12
Varicella (Infections and infestations) | 8 | 6 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Convulsion (Nervous system disorders) | 0 | 4 | 0
Headache (Nervous system disorders) | 2 | 5 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 5
Eczema (Skin and subcutaneous tissue disorders) | 4 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.